CLINICAL TRIAL: NCT02453776
Title: Precision Dosing Versus Conventional Dosing of Infliximab Maintenance Therapy: a Randomized Controlled Multicenter Study in Patients With IBD in Clinical Remission
Brief Title: Precision Dosing of Infliximab Versus Conventional Dosing of Infliximab
Acronym: PRECISION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, M. Lowenberg, dr, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2014_354
Record Dates: First submitted 2015-04-28; First posted 2015-05-27 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Inflammatory Bowel Disease
Keywords: Crohns Disease; Ulcerative Colitis; Infliximab; Sustained; Remission; Inflammatory bowel disease; IBD
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PRECISION dosing (Experimental): Infliximab may vary between 1-10 mg/kg and the interval between 4 and 12 weeks.
  Interventions: Drug: PRECISION dosing Infliximab
- Conventional dosing of Infliximab (No Intervention): Infliximab 5 mg/kg every 8 or 6 weeks

INTERVENTIONS:
Drug: PRECISION dosing Infliximab — Patients in the PRECISION dosing arm will recieve model based dosing, whereas proactive adjustments in treatment can be made by measuring the Infliximab concentration.
  Arms: PRECISION dosing

SUMMARY:
Infliximab (IFX) is highly effective in inducing and maintaining remission in patients with inflammatory bowel disease (IBD). However, a large proportion of patients will eventually lose response to IFX. Therefore, strategies to improve the outcome of maintenance treatment with IFX are required. Retrospective analyses suggest that adjusting IFX treatment in order to achieve IFX trough levels (TL) above a well-defined therapeutic threshold will improve the outcome of IFX treatment.

DETAILED DESCRIPTION:
Aim of this study is to investigate the efficacy of "precision dosing" IFX maintenance treatment in comparison with standard IFX maintenance treatment in IBD patients in clinical remission.

This study will be an open, randomized, controlled trial. Inclusion criteria: Patients aged ≥18 years with a diagnosis of Crohn's disease (CD) or ulcerative colitis (UC) based on endoscopy and pathology, receiving scheduled IFX therapy for ≥14 weeks, in clinical remission based on a Harvey Bradshaw Index (HBI) score ≤4 or a Partial Mayo (PM) score ≤2, for CD and UC, respectively. Exclusion criteria: Dilatation or resectional surgury in the past year and patients with a stoma/pouch.

Patients in the intervention arm will receive individualized treatment with variable IFX dosing AND/OR intervals guided by a Bayesian pharmacokinetic model, aiming to achieve an IFX TL of 3 µg/ml. Patients in the control group will continue to receive the same IFX treatment regimen that was given prior to inclusion without dose adaptation. In the control group, treatment adjustments will only be made in case of signs of active disease, in accordance to current routine care but these patients will be considered as failures to their treatment.

Primary endpoint: Proportion of patients with sustained clinical remission (based on HBI or PM). Secondary endpoints include: annual costs of IFX treatment per patient, total annual medical costs, side effects, (sustained) biochemical remission, adverse events, quality of life, IFX trough level and IFX antibodies (with an assay allowing presence of drug).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Participation will result in additional blood sampling, since IFX serum concentration will be measured every 8 weeks. All other laboratory tests can be considered as routine care. Patients in the intervention group with IFX TLs >3 will receive treatment de-escalation (interval elongation and/or dose reduction) as indicated by the Baysian model. Current evidence indicates that an IFX TL of 3 suffices. Patients in the intervention group with TLs <3 will receive treatment escalation (interval shortening and/or dose increase). We hypothesize that this will result in a higher chance of remaining in clinical remission.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CD or UC based on endoscopy and pathology
* 18 years or older
* Clinical remission, based on a Harvey Bradshaw Index (HBI) score ≤4 or a Partial Mayo (PM) score ≤2, for CD and UC
* Scheduled IFX maintenance treatment, regardless of interval/dosing

Exclusion Criteria:

- Dilatation or resectional surgery because of stenotic IBD in the past year

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Sustained clinical remission for the precision dosing group vs. the conventional IFX maintenance dosing group | 52 weeks
  Sustained clinical remission based on HBI (Crohn's disease) or PM score (Ulcerative Colitis)

SECONDARY OUTCOMES:
Cost of IFX treatment between the two groups | 52 weeks
  Comparing costs for treatment with IFX between the two groups
Proportion of patients with antibodies against IFX | 52 weeks
Quality of life | 52 weeks
  With a QoL questionnaire
Biochemical disease activity (CRP >5mg/L and fecal calprotectin ≥50% compared to baseline, to a value of >250 ug/g) | 26 weeks, 52 weeks
  A rise in fecal calprotectin of ≥50% compared to baseline, to a value of >250 ug/g and/or serum CRP of >5mg/L

CONTACTS AND LOCATIONS:
Overall Officials: G D'Haens, Study Director — Professor gastroenterology
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] Strik AS, Lowenberg M, Mould DR, Berends SE, Ponsioen CI, van den Brande JMH, Jansen JM, Hoekman DR, Brandse JF, Duijvestein M, Gecse KB, de Vries A, Mathot RA, D'Haens GR. Efficacy of dashboard driven dosing of infliximab in inflammatory bowel disease patients; a randomized controlled trial. Scand J Gastroenterol. 2021 Feb;56(2):145-154. doi: 10.1080/00365521.2020.1856405. Epub 2020 Dec 8. PMID 33290108